CLINICAL TRIAL: NCT05835674
Title: Multi-center Prospective Cohort Study CP-EDIT: Cerebral Palsy - Early Diagnosis and Intervention Trial
Brief Title: CP-EDIT: Cerebral Palsy - Early Diagnosis and Intervention Trial
Acronym: CP-EDIT
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other); Herlev Hospital (Other)
Responsible Party: Principal Investigator, Christina Høi-Hansen, Professor, MD, DMSc, Rigshospitalet, Denmark
Other Study IDs: H-22013292
Record Dates: First submitted 2023-03-31; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples. Whole genome sequencing will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort I: 500 participants screened by history and interview with parents to assess if they are to proceed to cohort II. This will be assessed by steering committee.
- Cohort II: Participants (n=300) who meet the inclusion criteria from Cohort I, is assessed at enrollment visit and will proceed to cohort III if they meet any two of the following criteria:
  1. Neuroimaging predictive of a motor disability
  2. GMA test with absent fidgety GMs at fidgety age
  3. HINE scores <57 at 3months or <60 at 6months or <63 at 9 months or < 66 at 12 months
  Infants will also be included if they meet both of the following criteria:
  1. Unilateral brain injury on neuroimaging predictive of CP
  2. Clinical signs of asymmetry
  Studies/objectives related to Cohort II
  1. Evaluation of MRI
  2. GMA implementation - To assess the feasibility of GMA in a multi-center Danish hospital setting.
  3. Prediction of CP - To determine the clinical utility of the MRI, HINE, HAI, and GMA to predict a confirmed diagnosis of CP at 24 months
  4. GMA/HINE/MRI vs. HAI - To compare diagnostic accuracy of HAI and GMA/HINE/MRI.
- Cohort III: Participants (n=160) will be included in cohort III if infants are considered CP or at high risk of CP Participants are followed at enrolment, and ages six, 12, 18 and 24 months. Blood sample for trio-whole genome sequencing is offered to participants with definite or high risk of CP.
  Studies/objectives related to Cohort III
  e) Evaluation of genetics f) GO-PLAY. To analyse the effect of the GO-PLAY intervention with early family-centred set-up for children with definite or high risk of CP.
  g) Parents perspective on intervention. To explore parents' perspectives on barriers and facilitators involved in early intervention.
  h) Parents perspectives of early diagnosis - To analyse interviews of parents' perspectives of gains and concerns when having an early diagnosis of high risk of CP.
  Interventions: Diagnostic Test: Early intervention program

INTERVENTIONS:
Diagnostic Test: Early intervention program — At enrollment visit: History and examination, MRI, evaluation of comorbidities, medication and genomic testing. HINE, GMA (if below 5 mo), AIMS, SHAI, PSS and DASS-21 questionnaire.
  At 6 mo visit: Examination and evaluation of comorbidities, medication and HINE and AIMS
  At 12 mo visit: Examination and evaluation of comorbidities, medication and HINE, AIMS, HAI, PSS and DASS-21 questionnaire.
  At 18 mo visit: Examination and evaluation of comorbidities, medication and HINE
  At 24 mo visit: Examination and evaluation of comorbidities, medication and HINE, PDMS-2, GMFM-66, BSID-IV-cog, MPOC-20 ,PSS, and DASS-21 questionnaire. GMFCS and Mini MACS if CP.
  Groups: Cohort III

SUMMARY:
Background. Early diagnosis of cerebral palsy is important as intervention becomes possible at a time where neuroplasticity is at the highest. Current mean age at diagnosis is 13 months in Denmark. Recent research has documented that implementation of an early-diagnosis set-up can lower diagnostic age of cerebral palsy. The aim of the current study is to show that the response to the early intervention program added to standard care is superior to standard care alone in a Danish multi-site setting in children from both a newborn and infant detectable risk pathway.

Methods The current study CP-EDIT (Early Diagnosis and Intervention Trial) with the GO-PLAY intervention included (Goal Oriented ParentaL supported home ActivitY program), aims at testing feasibility of an early diagnosis and intervention set-up in four paediatric centers. In a prospective cohort study design, we will consecutively include a total of 500 infants. We will systematically collect data at inclusion and follow a subset of participants with definite cerebral palsy or high risk of cerebral palsy until they are two years of age. The focus is on eight areas related to implementation and the perspective of the families: Early MRI; early genetic testing; implementation of the General Movements Assessment method; early prediction of cerebral palsy; comparative analysis of the Hand Assessment for Infants method and evaluation by Hammersmith Infant Neurological Examination, MRI, and the General Movements method; analysis of the GO-PLAY early intervention; parental perspective of early intervention; and parental perspective of having an early diagnosis.

Discussion Early screening for CP is increasingly possible and an interim diagnosis of "high risk of CP" is recommended but not currently used in our clinical care. There is a need to accelerate identification in mild or ambiguous cases to facilitate appropriate therapy early. The majority of studies on early diagnosis focus on identifying CP in infants below five months corrected age. Little is known about early diagnosis in the 50% of all CP cases that are discernible later in infancy, which is also addressed in this study. The study aims at improving care of patients with cerebral palsy even before they have the diagnosis established.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common cause of lifelong motor impairment in children and is defined by the Surveillance of Cerebral Palsy in Europe (SCPE) as "a group of permanent but not unchanging disorders of movement and/or posture and of motor function, which are due to a non-progressive interference, lesion, or abnormality of the developing/immature brain". An early diagnosis is important in order to start relevant intervention, when neuroplasticity is highest. Research suggests that early intervention programs have a positive influence on cognitive and motor outcomes and is a parental request.

In 2004, the Danish Cerebral Palsy Follow-up Program (CPOP) was introduced, with the aim of establishing a standardized follow-up program. The CPOP guarantees that children with CP are followed annually and aims to document, monitor, and improve the quality of health care for children with CP in Denmark. A previous Danish nationwide study from birth years 1995-2003 found that the median corrected diagnostic age of Danish children with CP was 11 months based on first mention in the patient journal. In an novel analysis we have found that for children with CP in birth years 2010-2013 the diagnostic age was 13 months based on first registered diagnosis. The best predictive tools for early diagnosis of CP has been found to be the Prechtl Qualitative Assessment of General Movements (GMA), Hammersmith Infant Neurological Examination (HINE) and cerebral MRI. These tools can be used to diagnose CP before the corrected age of five months. The method Hand Assessment for Infants (HAI) has in recent publications been found promising to complement these tests, but little evidence on HAI has been published. Feasibility of an early-diagnosis set-up of a systematic approach with neurological assessment, GMA/HINE and neuroimaging has been evaluated in several studies, but not yet in Denmark and not in a setting where both the newborn- and infant-detectable risk pathways were included. Neonates may have obvious risk factors at birth/in the neonatal period, but in the present study infants with findings suggesting CP emerging in the first year of life are also included.

For more than 80% of children with CP neuroimaging performed with MRI is abnormal. It has been recommended for many years to use MRI while diagnosing CP. A review from 2007 showed that 86% of the MRIs performed on children with CP were abnormal and for the majority gave clues to the pathogenesis of CP. In a previous Australian study of children with CP specific MRI patterns varied depending on parity, gestational age, level of neonatal care, Apgar score and time to established respiration. Diagnostic MRI of newborns and infants with suspected brain damage are today based on structural images with the focus on identifying major structural brain pathology, such as periventricular leukomalacia or white matter damage. However, advanced research MRI-sequences can be sensitive to detect brain damage and may provide important biological information about myelination, microstructure, and connectivity of the white matter fibre tracts, as well as the metabolic profile, including markers of neuronal integrity and glial markers, of the brain tissue. MRI will be offered earlier than regular clinical practice for participants in this research project and for a subset of patients repeat MRI will be possible.

Many gene variants may play a role in the development of CP. Previous research with genetic testing has shown that genetic aetiology, while often seen in children with no previous gestational or neonatal risk factor, is not limited to this group nor those with other neurodevelopmental comorbidities such as epilepsy or intellectual disability. One study has suggested an association between CP and genes that hinder early brain development and also predispose to susceptibility to environmental risk factors. The cause for the various CP types, including the most prevalent spastic subtype and the rare ataxic or dyskinetic CP, are different. In some cases, the cause is obvious, such as asphyxia during labour, cerebral bleeding, or infection, but in many cases the cause is unknown. However, in an increasing number of patients it is now possible to identify the underlying cause, since it has become clear that several treatable metabolic and genetic diseases such as dopa-responsive dystonia may be misdiagnosed as CP. Identifying the cause makes it possible to provide genetic counselling and direct specific treatment, e.g., with nutrient-specific diets or medications, which can interrupt disease progression and hinder further injury. In the current study extensive genetic testing with whole genome sequencing will be performed in participants with definite CP or high risk of CP.

Receiving an early diagnosis of CP or high risk of CP is a parent priority and both parents and care providers agree that early access to interventions is important for the child. Parents of children with CP may experience high stress levels, depression, and chronic sorrow symptoms. Intensive home-based approaches addressing cognitive and motor improvement increasingly involve parents as treatment providers, supervised by therapists. This can lead to both a positive parental outcome such as motivation, knowledge, and increased competences, as well as negative outcomes, because parents may be overwhelmed by the burden of responsibility and the feeling of insufficiency and lack of confidence.

The current study CP-EDIT (Early Diagnosis and Intervention Trial) with the GO-PLAY intervention included ( Goal Oriented ParentaL supported home ActivitY program, that will be registered separately at ClinTrials), aims at testing feasibility of an early diagnosis and intervention set-up in four neuropaediatric centers in Denmark with focus on eight areas related to implementation and the perspective of the families: Early MRI, early genetic testing, implementation of the GMA method, early prediction of CP, comparative analysis of the HAI and HINE, MRI, and GMA methods, analysis of the GO-PLAY early intervention, and parental perspective of intervention and early diagnosis.

ELIGIBILITY:
Inclusion Criteria:

Group A: 'Newborn-detectable risk-pathway'

* Preterm birth with gestational age below 32 or birth weight below 1500 g and clinical concern
* Moderate to severe brain injury (Papile grade 3 to 4 intraventricular haemorrhage, cystic periventricular leukomalacia, neonatal stroke, term hypoxic-ischaemic encephalopathy (≥35 weeks gestation at birth) or other significant neurological condition)
* History (e.g. neonatal seizures, Extra Corporal Membrane Oxygenation, meningitis, kernicterus, severe hypoglycemia) or neurological risk factors (brain malformation, increased tone)
* Parental concern and one of the factors above

Group B: 'Infant detectable risk-pathway'

* Inability to sit independently by age 9 months
* Hand function asymmetry or crawl asymmetry
* Inability to take weight through the plantar surface of the feet
* History (as above) or neurological risk factors
* Parental concern and one of the factors above

Exclusion Criteria:

* 1) Infants with progressive or neurodegenerative disorders or genetic disorders not associated with CP, 2) Infants with other disability diagnoses e.g. Down Syndrome.

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants below 12 months of age with risk of cerebral palsy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
MRI | MRI at enrollment in cohort II
  MRI scans will be described clinically by radiologists at the participating hospitals. The findings will be categorised according to SCPE criteria (Surveillance of Cerebral Palsy in Europe). In participants where ultrasound or CT scanning of the patients have already been performed as part of clinical follow-up, the results will be gathered, and additional MRI may be optional. Repeat MRI at ages 12 and 24 months will be optional for participants in cohort III as part of the complementary NIBS-CP project (NeuroImaging of Babies during natural Sleep to assess typical development and Cerebral Palsy), which may provide important biological information about myelination, microstructure, and connectivity of the white matter fibre tracts, as well as the metabolic profile, including markers of neuronal integrity and glial markers, of the brain tissue
Whole genome sequencing | Genetics at enrollment in cohort III
  Blood samples will be obtained from participants with definite or high risk of CP (n=160) upon inclusion in CP-EDIT cohort III after informed, written consent has been obtained by the parents. The parents will also be asked to provide a blood sample and written consent for genome sequencing (trio-analysis). A clinical geneticist and clinical laboratory geneticist will perform the data analysis and result interpretation. Results will be categorised as either: I) Pathogenic CP-explaining variant, II) Likely pathogenic CP-explaining variant, III) Variant of uncertain significance, IV) Likely benign variant, V) Benign variants (according to the ACMG guidelines) and VI) Pathogenic variant, non-CP disease. Only data from the proband will undergo a full analysis. De novo variants in gene with no known clinical association may be submitted to GeneMatcher.
Hammersmith Infant Neurological Examination (HINE) | At enrollment visit
  The HINE is a standardized neurological examination for infants aged 3-24 months. It includes three sections: 1) Neurological Examination - Assessment of cranial nerve function, posture, movements, tone, reflexes and reactions 2) Motor Milestones - head control, sitting, grasping, rolling, crawling, standing and walking and 3) State of Behavior - consciousness, emotional state and social orientation. The HINE global score ranges from a minimum of 0 to a maximum score of 78. A score < 73 indicates high risk of CP and < 40 indicates abnormal outcome, usually CP. HINE cut off scores for high risk infants indicating CP are: score < 57 at 3 months, <60 at 6 months, < 63 at 9 months and, < 66 at 12 months. The HINE asymmetry-score, also provides insight into CP topography (unilateral vs bilateral) and CP motor severity (ambulant vs non-ambulant, GMFCS I-III vs IV-V). The HINE is performed by a neuro pediatrician or physiotherapist.
General Movement Assessment (GMA) | At enrollment visit if < 5 months of corrected age
  GMA is an observation that evaluates the quality of an infant's early spontaneous movement patterns. GMA is categorised in writhing movements (from preterm until 6-9 weeks post term age) and fidgety movements (from 9 to 20 weeks post term age). Absent fidgety movements (FM) at 3 months post-term age is highly predictive of CP in 'high-risk' infants and may be a marker for other adverse neurodevelopmental outcomes. FMs are classified as follows: Normal, defined as circular movements of small amplitude, moderate speed, and variable acceleration of neck, trunk, and limbs in all directions. Abnormal FMs: (a) absent, when normal FMs are never observed from age 9 to 20 weeks post term age; (b) sporadic , when FMs can be detected but less than 3 sec. (c) exaggerated, when FMs are of large amplitude, high speed, and jerkiness are seen.
Screening Hand Assessment for Infants (SHAI) | At enrollment visit
  SHAI is developed to facilitate screening for risk of unilateral CP in infants aged 3-12 month at risk of CP. The sHAI measures the manual actions performed with each hand separately, test procedure comprises a semi-structured video-recorded play session lasting 5 min, with assessment of 6 unimanual items (including quality of holding, grasping from easy position, object location, finger movements and quality of movement). All items are scored on a three-point rating scale (0-2) and the scores of the unimanual items are summed to the Each Hand Sum score (EaHS) with a range of 0-12 raw scores. The EaHS of the better functioning hand and the lesser functioning hand is used to calculate an asymmetry index (0-100) where a higher percentage indicates a larger asymmetry.
Clinical assessment of CP diagnosis | at 24 months corrected age
  Definitely CP' encompasses participants that fulfil SCPE CP clinical criteria and guided by fulfilling the following: 4/5 for children <5 months, and 3/4 for children ≥ 5 months of the following at screening.
  1. Delayed motor development without signs of neuromuscular disease (floppy infant, absent reflexes)
  2. GMA test with absent fidgety GMs at fidgety age
  3. HINE scores <57 at 3months or <60 at 6months or <63 at 9 months or <66 at 12 months
  4. MRI or ultrasound of brain with a lesion in one or more of the following structures: sensori-motor cortex, basal ganglia, posterior limb of the internal capsule, pyramidal tracts
  5. Focal neurological symptoms (hyperreflexia, clonus, dystonia, ataxia, intention tremor) or clinical signs of asymmetry

SECONDARY OUTCOMES:
Motor function - The Gross Motor Function Classification System - Expanded & Revised (GMFCS - E&R) | at 24 months corrected age
  GMFCS - E&R is a 5-level classification system that describes the gross motor function of children and youth with CP based on their self-initiated movement with particular emphasis on sitting, walking, and wheeled mobility. Distinctions between levels are based on functional abilities, the need for assistive technology, including hand-held mobility devices (walkers, crutches, or canes) or wheeled mobility, and to a much lesser extent, quality of movement. The GMFCS - E&R contains 5 age bands (under 2 years, 2-4 years, 4-6 years, 6-12 years, and 12-18 years) and is categorized into five levels from walking without limitation (level I) to non-ambulatory function (levels IV and V)
Motor function - The Mini-Manual Ability Classification System (Mini-MACS) | at 24 months corrected age
  Mini-MACS describes how children with CP aged 1-4 years use their hands when handling objects in daily activities. Ability is ranked on five levels based on the children's self-initiated ability and their need for assistance or adaptation when handling objects. The five levels are categorized from able to handle objects easily and successfully (level 1) to does not handle objects and has severely limited ability to perform even simple actions (level 5). Mini-MACS is a functional description that can be used as a complement to the supposed diagnose of CP and its subtypes.

OTHER OUTCOMES:
Motor Optimality Score - Revised (MOS-R) | At enrollment visit if < 5 months of age
  MOS-R is the detailed GMA for 3-5-month-old infants. The MOS-R comprises the following five subcategories: (1) Quality of fidgety; (2) Observed movement patterns; (3) age-adequate movements (4) Observed postural patterns and (5) movement character. The MOS score ranges from a minimum of 5 to a maximum score of 28. An MOS ranging from 25 to 28 is considered to be optimal; scores from 20 to 24 are mildly reduced and an MOS below 20 requires intervention. A score below 9 indicates a very high risk for neurodevelopmental disabilities, especially for non-ambulatory CP.
Alberta Infant Motor Scale (AIMS) | At enrollment, six and 12 months corrected age
  AIMS is an observational assessment scale constructed to measure gross motor maturation in infants from birth through independent walking. 58 items are generated and organized into four positions: prone, supine, sitting and standing. Each item describes three aspects of motor performance weight-bearing, posture and antigravity movements. The overall score ranges from a minimum of 0 to a maximum of 58.
Peabody Developmental Motor Scales - Second edition (PDMS-2) | at 24 months corrected age
  PDMS-2 is a standardized, norm-referenced measure used to evaluate the gross and fine motor development of children aged birth to 6 years. The gross motor component is comprised of four subtests: reflexes (raw score range 0-16), stationary (raw score range 0-60), locomotion (raw score range 0-178) and object manipulation (raw score range 0-48). Two subtests, grasping (raw score range 0-52) and visual-motor integration (raw score range 0-144), form the fine motor component. The total Motor Quotient (TMQ) is formed by a combination of the results of the gross and fine motor subtests. The PDMS-2 TMQ range from 90-165 (indicating average or above average age-normed motor abilities) to 89-35 (indicating below average to very poor age-normed motor abilities).
Gross Motor Function Measure (GMFM-66) | at 24 months corrected age
  GMFM-66 is a criterion-referenced tool designed and evaluated to measure changes in gross motor function over time or with intervention in children with CP. It consists of 5 dimensions rolling, sitting, walking, running, and jumping. The 66 items are organized in increasing difficulty order from 0 (low capacity) to 100 (high capacity) along an interval scale. Each item is scored on a four-point Likert scale (0-3). It can be used from 5 months of age, and a 5- year-old typically developing child is expected to achieve a score of 100.
Bayley Scales of Infant and Toddler Development 4-cognitive | at 24 months corrected age
  BSID-4 is a standardized and norm-referenced assessment, which measures the cognitive, motor, language and social-emotional development of infants and toddlers aged 0-3. Raw scores of successfully completed items are converted to scale scores and to composite scores. These scores are used to determine the child's performance compared with norms taken from typically developing children of the same age.
HINE | at visit six, 12, 18, and 24 months corrected age
  The HINE is a standardized neurological examination for infants aged 3-24 months. It includes three sections: 1) Neurological Examination - Assessment of cranial nerve function, posture, movements, tone, reflexes and reactions 2) Motor Milestones - head control, sitting, grasping, rolling, crawling, standing and walking and 3) State of Behavior - consciousness, emotional state and social orientation. The HINE global score ranges from a minimum of 0 to a maximum score of 78. A score < 73 indicates high risk of CP and < 40 indicates abnormal outcome, usually CP. HINE cut off scores for high risk infants indicating CP are: score < 57 at 3 months, <60 at 6 months, < 63 at 9 months and, < 66 at 12 months. The HINE asymmetry-score, also provides insight into CP topography (unilateral vs bilateral) and CP motor severity (ambulant vs non-ambulant, GMFCS I-III vs IV-V).
Hand Assessment in Infants (HAI) | at 12 months corrected age
  HAI is an assessment developed for infants at risk of developing CP in the age range 3-12 months. The test procedure comprises a semi-structured video-recorded play session lasting 10- 15 min. A test kit of toys is presented to the infant to encourage and elicit exploration, making a wide range of a unilateral and bilateral hand movements observable. The HAI measures the degree and quality of goal directed actions performed with each hand separately as well as both hands together. It provides a separate score for each hand (Each Hand Sum Score 0-24), a score for both hands (Both Hands Sum Score 0-58), an asymmetry index in % illustrating possible asymmetric hand use as well as criterion referenced measure of general upper limb ability (HAI-units 0-100)
The Depression Anxiety Stress Scales (DASS-21) | at enrollment visit, and 12, 24 months corrected age
  DASS-21 is an adult self-report designed to measure the emotional states of depression, anxiety and stress. It is a 21-item questionnaire and will be used to measure parent emotional well-being
The Parental stress scale (PSS) | at enrollment visit, and 12 and 24 months corrected age
  PSS is an 18-item questionnaire assessing parents' feelings about their parenting role, exploring both positive (emotional benefits, personal development) and negative aspects (demands on resources, feelings of stress) of parenthood. The overall score ranges from a minimum of 18 to a maximum of 90
The Ages & Stages Questionnaire (ASQ-3) | at 24 months corrected age
  ASQ-2 pinpoints developmental progress in children between the age of one month to 5 ½ years. It has a parent-centric approach and is used as a developmental screener
The Measure of Processes of Care 20 (MPOC-20) | at 24 months corrected age
  MPOC-20 is a self-report measure of parents' perceptions of the extent to which the health services they and their child(ren) receive are family-centered. The 20 items consist of 5 domains; enabling and partnership, providing general information, providing specific information about the child, respectful and supportive service, and coordinated and comprehensive care.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Hoei-Hansen, professor, Study Chair — Department of Paediatrics, University Hospital Rigshospitalet, Denmark
Locations (4):
- Denmark (4):
  - University Hospital Aalborg, Aalborg
  - University Hospital Aarhus, Aarhus
  - University Hospital Herlev, Herlev
  - University Hospital Rigshospitalet, Dept. Paediatrics, Copenhagen, Østerbro

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing options are being explored.